CLINICAL TRIAL: NCT02674815
Title: Preoperative High Intensity Interval Training in Patients Scheduled for Colorectal and Thoracic Surgery: The PHIIT Trial
Brief Title: Preoperative High Intensity Interval Training: The PHIIT Trial
Acronym: PHIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Jonathan Moran, Mr, University of Dublin, Trinity College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRFSJ0086
Record Dates: First submitted 2016-01-26; First posted 2016-02-05 (Estimated); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Neoplasms; Lung Neoplasms
Keywords: Exercise; Preoperative; High Intensity Interval Training; Colorectal; Thoracic; Postoperative
MeSH Terms: conditions — Colorectal Neoplasms; Lung Neoplasms; Motor Activity

ARMS (1):
- Intervention (Experimental): Patients within this arm will perform two weeks of high intensity interval training prior to colorectal/thoracic surgery. Exercise intensity will be 100% of the peak power output (PPO) during maximal cardiopulmonary exercise testing. Patients will exercise for 15 seconds at 100% PPO and rest for 15 seconds (passive) for 30 minutes or until exhaustion. This will be performed 5 days a week for 2 weeks.
  Interventions: Other: High Intensity Interval Training Exercise programme

INTERVENTIONS:
Other: High Intensity Interval Training Exercise programme — High intensity interval training (HIIT) requires participants to exercise at high levels of VO2peak (≥80% VO2peak). Participants exercise for short periods (e.g. 15-30 seconds) followed by periods of rest (active or passive) and typically continue this pattern for a set time period or until exhaustion.
  Other Names: HIIT

SUMMARY:
Colorectal and thoracic surgical patients are susceptible to poor postoperative outcome including complications, mortality and increased length of stay. Preoperative physical fitness is protective against poor postoperative outcome in intra-abdominal and thoracic surgery.

The current colorectal/thoracic pathway from diagnosis to surgery is about 2 weeks and therefore interventions of longer duration are not feasible. Clinicians may be presented with a difficult choice in delaying surgery to perform prehab or cancel the pre-op intervention.

To create greater improvements in aerobic fitness, participants are required to exercise at high levels of VO2peak (e.g. ≥80% VO2peak). High intensity interval training (HIIT) requires participants to exercise at high levels of VO2peak (≥80% VO2peak) for short periods (e.g. 15 seconds) followed by a recovery (active or passive) and typically continue this pattern for 30 minutes or until exhaustion.

HIIT programmes are safe and a recent meta-analysis noted that HIIT produced a more pronounced incremental gain in participants' mean VO2peak when compared with continuous moderate intensity exercise (+1.78mL/kg/min, 95% CI: 0.45-3.11).

HITT has not been investigated as a preoperative intervention to either optimize fitness prior to surgery or reduce post-surgical complications. Preoperative HIIT is an intense intervention which will require significant participant adherence. The safety, cost and clinical application of such a programme needs to be performed. This feasibility study aims to assess the ability of HIIT to improve aerobic fitness two weeks prior to surgery and determine its feasibility.

DETAILED DESCRIPTION:
Colorectal and thoracic surgical patients are susceptible to poor postoperative outcome. In colorectal surgery the rate of post-op complications is between 15-20% and the rate of 30 day mortality is 2.3%. Thoracic surgery also carries significant risk, 30 day mortality is 2.2% while the rate of post-op complications is 29.3%. Poor postoperative outcome significantly affects the patients recovery and increases hospital costs. Reducing postoperative risk therefore conveys significant benefit to the patient and the hospital.

Preoperative physical fitness is predictive of postoperative outcome in intra-abdominal and thoracic surgery. In a systematic review of 6 studies preoperative exercise interventions improved pre-op physical fitness in patients undergoing abdominal surgery, however it is unclear if this translates into an improvement in postoperative outcome.

An updated systematic review and meta-analysis was performed on the effects of pre-habilitation on postoperative outcome. While the results demonstrated that preoperative exercise interventions of 4-6 week duration reduced post-op complications a significant amount of work is still to be performed in this area.

The current colorectal/thoracic pathway from diagnosis to surgery is about 2 weeks and therefore interventions of longer duration are not feasible. Clinicians may be presented with a difficult choice in delaying surgery to perform prehab or cancel the pre-op intervention.

To create greater improvements in aerobic fitness, participants are required to exercise at high levels of VO2peak (e.g. ≥80% VO2peak). High intensity interval training (HIIT) requires participants to exercise at high levels of VO2peak (≥80% VO2peak). Participants exercise for short periods (15 seconds) followed by 15 seconds of rest and typically continue this pattern for 30 minutes or until exhaustion.

A recent review reported HIIT programmes to be safe in individuals with coronary artery disease and stable heart failure. In agreement with this paper a recent meta-analysis noted that HIIT produced a more pronounced incremental gain in participants' mean VO2peak when compared with continuous moderate intensity exercise There are a number of factors to take into account when designing a HIIT programme e.g. duration and intensity of exercise phase and type of recovery period (active vs. passive). Two papers compared a selection of HIIT protocols for safety and time at a high percentage of VO2peak (≥ 80% VO2peak). Protocols with rest periods (passive recovery) allowed patients to exercise for longer and had lower perceived difficulties. In one study of 20 patients with CAD, HITT was prescribed with 15s exercise and passive recovery intervals at 100% Peak Power Output (PPO) or Maximal Aerobic Power (MAP) with no adverse events. PPO or MAP is the power of the last completed stage during a maximal exercise test (watts). This intervention had the highest duration above 80% VO2peak (819s) and a high completion rate of 63%. This protocol was chosen for this study.

HITT has not been investigated as a preoperative intervention to either optimize fitness prior to surgery or reduce postsurgical complications. Preoperative HIIT is an intense intervention which will require significant participant adherence. The safety, cost and clinical application of such a programme needs to be performed. This feasibility study aims to assess the ability of HIIT to improve aerobic fitness two weeks prior to surgery and determine its feasibility.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for colorectal or thoracic surgery
2. Able to give informed consent
3. Ability to understand English

Exclusion Criteria:

* Acute myocardial infarction
* Unstable angina
* Uncontrolled arrhythmias causing symptoms or hemodynamic compromise
* Syncope
* Active endocarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolous or pulmonary infarction
* Thrombosis of lower extremities
* Suspected dissecting aneurysm
* Uncontrolled asthma
* Pulmonary edema
* Room air desaturation at rest ≤85%
* Respiratory failure
* Acute noncardiopulmonary disorder that may affect exercise performance or be aggravated by exercise (i.e. infection, renal failure, thyrotoxicosis)
* Cognitive impairment leading to inability to cooperate
* Left main coronary stenosis or equivalent
* Moderate stenotic valvular heart disease
* Severe untreated arterial hypertension at rest (>200 mmHg systolic, >120 mmHg diastolic)
* Tachyarrhythmias or bradyarrhythmias
* High-degree atrioventricular block
* Hypertrophic cardiomyopathy
* Significant pulmonary hypertension
* Pregnancy
* Electrolyte abnormalities
* Orthopaedic impairment that compromises exercise performance
* Individuals with pacemakers or defibrillators
* Epilepsy
* Past history or MRI evidence of brain damage, including significant trauma, stroke, transient ischaemic attack (TIA), hydrocephalus, mental retardation, or serious neurological disorder
* Non resectable disease
* Emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2016-02; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cost | 6 months
  The cost of the programme will be recorded. Expected costs include, parking, room rental charges, equipment rates, employee rates.
Adherence/Compliance | 6 months
  The adherence rates will be measured by recording the number of appointments each participant attends.
  The number of missed sessions per participant and the reasons for missing sessions will be recorded and reported. If a participant misses an exercise sessions they will be contacted by the research team to determine the reason and to reschedule the class for later that day if possible. If a participant misses more than 50% of total exercise sessions in the absence of a defined reason (acute illness or scheduled holiday), it will be recorded as a protocol violation.
Incidence of Adverse Events | 6 months
  Adverse events will be assessed at every clinic visit and the following details recorded: type, incidence, severity, timing, seriousness, and relatedness to a) disease and b) the intervention.
Satisfaction/Acceptability | 6 months
  Self-administered questionnaire on completion of programme will be administered. Participants will also be asked to highlight what they liked and didn't like about the programme and any suggestions for change.
Withdrawal of participants | 6 months
  Participants are free to withdraw from the trial at any stage without providing a reason and without consequence. This information will be stated in the participant information leaflet. Participants can inform the research team at their local site of their decision to withdraw. If a participant withdraws from the study, any data collected on them up to that point in the study will go forward for study analysis. This information will be stated in the participant information leaflet. If a participant withdraws from the intervention, but provides consent to complete subsequent follow-up measurements they will continue to attend study assessments and data will be used for intention-to-treat analysis. Participants will be asked for their reason to withdrawing consent, participants are not required to give a reason. Reasons for stopping the intervention will be recorded and reported
Protocol deviations/Adaptations | 6 months
  The following deviations will be recorded and reported.
  • Changes to exercise protocol (e.g. reduction in number of sessions, change in % PPO performed during exercise session)
Compliance | 6 months
  Compliance will be measured in the percentage of exercise sessions attended and successfully completed.

SECONDARY OUTCOMES:
Postoperative mortality | Up to day 30 post-op
  Postoperative mortality will be recorded until day 30 post-op.
Changes in Aerobic Capacity | 6 months
  Participants will perform a maximal CPET prior to beginning of intervention to establish baseline aerobic fitness. Upon completion of the intervention, prior to surgery, participants will repeat the maximal CPET.
Length of stay | 6 months
  Length of stay will include general hospital stay from time of operation to discharge, ICU/HDU admission rates and length of stay as well as readmission rates.
Postoperative complications assessed using the Postoperative Morbidity Survey | Up to 7 days post-op
  Postoperative morbidity will be assessed using the postoperative morbidity survey (POMS) (type and number of complications on a specific day). POMS will be performed on Day 3, 5, 6 and 7.
Readmission rates | 6 months
  The amount of readmission's to hospital due to surgery related reasons.
ICU/HDU admission rates | 6 months
  The amount of admissions to the Intensive Care Unit/High Dependency Unit due to surgery related reasons
ICU/HDU length of stay | 6 months
  The amount of time (recorded in days) a patient spends in ICU/HDU due to surgery
Clavien-Dindo Classification Sore | 6 months
  The most severe complication experienced by a patient will be assessed and recorded using the Clavien-Dindo Classification Score

CONTACTS AND LOCATIONS:
Locations (1):
- St. James's Hospital, Dublin, Ireland